CLINICAL TRIAL: NCT01709136
Title: Pharmacokinetics of Sirolimus and Tacrolimus in Liver Transplant Recipients With Early Nephrotoxicity and/or Hypertension Due to Tacrolimus
Brief Title: Pharmacokinetics of Sirolimus and Tacrolimus in Liver Transplant Recipients With Tacrolimus Toxicity
Acronym: Sirolimus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sirolimus usage discontinued since black box warning
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rakesh Sindhi, Professor of Surgery, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07100379
Record Dates: First submitted 2010-06-29; First posted 2012-10-17 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental)
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the Children's Hospital of Pittsburgh's Pediatric Clinical and Translational Research Center (PCTRC) - See more at: http://www.chp.edu/research/our-facilities/pctrc, and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab. This phase can either be performed immediately after the 12-hour iothalamate GFR evaluation, or a few days later at the convenience of the subject.
  Other Names: Sirolimus (Rapamycin); Tacrolimus (FK506)

SUMMARY:
Pharmacokinetics of Tacrolimus and Sirolimus alone and in combination in liver transplant recipients.

DETAILED DESCRIPTION:
Liver transplant patients receiving tacrolimus, and who experience side effects such as hypertension and renal dysfunction, will be converted to sirolimus with low-dose tacrolimus, or Tacrolimus withdrawal. This study will evaluate allograft function by serial clinical lab testing, the pharmacokinetics of sirolimus and tacrolimus, the glomerular filtration rate (GFR) and the potential side effect of sirolimus, such as marrow suppression and hyperlipidemia. Two pharmacokinetic evaluations are planned: once around the third post-transplant month and another one at about 12 months. Expected outcomes are, a better understanding of sirolimus pharmacokinetic parameters over time in pediatric/adult liver recipients and early efficacy and safety data of the sirolimus as a non-nephrotoxic alternative to tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of primary liver (cadaver/liver, whole/segmental) transplants 5- 30 years old.
* Rejection-free post-transplant course for at least 3 months
* Renal dysfunction (15% decrease in age-adjusted calculated creatinine clearance)
* Hypertension requiring anti-hypertensive mediations.
* Informed consent.
* Weight ≥15 kg.

Exclusion Criteria:

* Rejection or infections within 3 months of enrollment.
* Intent to continue TAC
* Active participation in ongoing studies of immunosuppressive agents.
* Lack of informed consent.
* Pregnant or breast feeding
* HIV positive

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sindhi, Principal Investigator — UPitt

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Sirolimus: Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the Children's Hospital of Pittsburgh Pediatric Clinical and Translational Research Center (PCTRC) - See more at: http://www.chp.edu/research/our-facilities/pctrc, and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab. This phase can either be performed immediately after the 12-hour iothalamate Glomerular Filtration Rate (GFR) evaluation, or a few days later at the convenience of the subject.
Period: Overall Study
Arm/Group | Sirolimus
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sirolimus: Sirolimus: Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the PCTRC , and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab. This phase can either be performed immediately after the 12-hour iothalamate GFR evaluation, or a few days later at the convenience of the subject.
Arm/Group | Sirolimus
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Secondary Outcome: PK Parameters for Tacrolimus and Sirolimus
Description: pharmacokinetics (PK) of SRL after a single dose and after steady state has been achieved; and the pharmacokinetics of tacrolimus once at steady state
Time Frame: 12 months
Population: We were able to preform 3 pharmacokinetics (PK) profiles, one in each of three patients enrolled. However, due to emerging data and blackbox warnings from FDA suggesting that use of Sirolimus in liver transplant recipients be circumspect (risk of thrombosis and death), the study was terminated early and data analysis was not able to be completed.
Groups:
- Sirolimus: Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the PCTRC , and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab.
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

2. Secondary Outcome: SRL Can Substitute TAC
Description: Whether Sirolimus can substitute Tacrolimus in the stable post-transplant state, without compromising allograft function
Time Frame: 12 months
Population: Due to FDA blackbox warnings (6/11/09) about Sirolimus in liver transplant recipients (risk of thrombosis and death), the study was terminated early. Due to the early termination of this study and small number of subjects enrolled (3), data analysis was not able to be completed.
Groups:
- Sirolimus: Sirolimus: Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the PCTRC , and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab..
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

3. Primary Outcome: Early and Late Pharmacokinetics of Sirolimus (SRL)
Description: To evaluate early and late pharmacokinetics of Sirolimus (SRL) , and safety and efficacy of conversion from tacrolimus (TAC) to sirolimus in liver transplant recipients who have been stable for at least 3 months, and who have early nephrotoxicity and/or hypertension due to use of tacrolimus.
Time Frame: 1 year
Population: Three pharmacokinetics (PK) profiles were performed, one in each of three patients who were enrolled. However, due to FDA blackbox warnings (6/11/2009) about Sirolimus in liver transplant recipients be circumspect (risk of thrombosis and death), the study was terminated early and data analysis was not able to be completed.
Groups:
- Sirolimus: Single dose SRL pharmacokinetics and TAC steady state pharmacokinetics: This phase is applicable to both sets of patients: those with nephrotoxicity and those with hypertension. Patients will receive a single dose of SRL of 2 mg/m2. Blood sampling will be performed over a 24 hour stay in the PCTRC, and the sampling for 48 hour and 72 hour PK studies can be done at the outpatient lab.
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

4. Secondary Outcome: SRL Prevent TAC-related Side Effects
Description: Whether SRL can prevent or minimize progression of selected TAC-related side-effects such as renal dysfunction as measured by clearance of iothalamate (Glomerular filtration rate < 80 mL/min/1.73 m2) and hypertension (blood pressure > 140/90 mm Hg)
Time Frame: 1 year
Population: Due to FDA blackbox warnings from FDA (6/11/2009) about Sirolimus in liver transplant recipients (risk of thrombosis and death), the study was terminated early and data analysis was not able to be completed.
Arm/Group | Sirolimus
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: There have been no adverse events or unanticipated events during the course of this study.
Arm/Group | Sirolimus
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Complete follow-up failed, due to early study termination as a result of FDA black box warning (6/11/2009) about Sirolimus in liver transplant recipients (risk of thrombosis and death).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes